CLINICAL TRIAL: NCT01548859
Title: Comparison of the Effects of Sevoflurane and Midazolam Used for the Maintenance of Anaesthesia on the Levels of Postoperative Cardiac Troponin I in Pediatric Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Huseyin Utku YILDIRIM, Anaesthesiology Resident, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KA 11/60
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Myocardial Injury; Anaesthetic Preconditioning
Keywords: Myocardial protection; Myocardial injury; Anaesthetic preconditioning; Pediatric cardiac surgery; Troponin I; Sevoflurane; Midazolam
MeSH Terms: interventions — Midazolam; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Active Comparator): Used for maintenance anaesthesia (0.2 mg/kg/saat continuous infusion)
  Interventions: Drug: Midazolam
- Sevoflurane (Active Comparator): Used for the maintenance for anaesthesia (% 0.5-8 end tidal concentration)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Midazolam — 0.2 mg/kg/saat continuous infusion of midazolam received during anaesthesia
  Arms: Midazolam
Drug: Sevoflurane — end tidal concentration of % 0,5-8
  Arms: Sevoflurane

SUMMARY:
The purpose of this study is to compare two different anaesthetic agent effect on postoperative Troponin I levels in pediatric cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective pediatric surgery
* Patients written informed consent for study participation

Exclusion Criteria:

* Redo surgery
* History of myocarditis
* Renal failure
* Pulmonary embolism
* Hypothyroidism

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
myocardial protective effect of sevoflurane | postoperative 48 hours
  Postoperative troponin I levels

SECONDARY OUTCOMES:
Hemodynamic and respiratory data | Postoperative 48 hours
  Arterial pressure, heart rate, blood gas analysis, extubation time,

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Faculty of Medicine, Ankara, Çankaya, Turkey (Türkiye)